CLINICAL TRIAL: NCT05977582
Title: Prevention Program for Eating Disorders Applied to College Students Using a Virtual Platform. Spanish Validation of the eBodyProject
Brief Title: Online Prevention Program for Eating Disorders Applied to College Students. Spanish Validation of the eBodyProject
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: University of Burgos (Unknown)
Responsible Party: Principal Investigator, Carmen Varela, PhD, Researcher and Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IR15/2023
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Eating Disorders
Keywords: Prevention; College women; Thin-ideal internalization
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spanish Version eBodyProject (Experimental): The Spanish adaptation of the eBodyProject program will be modified (Stice et al., 2012b). This program consists of 4 modules adapted from the most recent version of the original program The Body Project, presented by the original authors who have given their consent and suggestions for the realization of the Spanish version.
  The activities proposed through the different modules will be in written format or behavioral activities aimed at criticizing the ideal of feminine beauty imposed by today's society and promoting self-acceptance.
  Interventions: Behavioral: Spanish version eBodyProject
- Psychoeducational Prevention Program (Active Comparator): Participants in this group will receive a weekly newsletter with information about the beauty ideal, the costs of pursuing it, and tips for resisting the pressure to pursue this ideal, as well as tips for managing the emotions associated with it. However, they will not have to perform exercises related to this information, a psychoeducational intervention. Once the study is finished, these participants will receive an email again in case they are interested in taking part in the eBodyProject prevention program.
  Interventions: Behavioral: Psychoeducationa Prevention Program

INTERVENTIONS:
Behavioral: Spanish version eBodyProject — The Spanish adaptation of the eBodyProject program will be modified (Stice et al., 2012b). This program consists of 4 modules adapted from the most recent version of the original program The Body Project, presented by the original authors who have given their consent and suggestions for the realization of the Spanish version.
  The activities proposed through the different modules will be in written format or behavioral activities aimed at criticizing the ideal of feminine beauty imposed by today's society and promoting self-acceptance.
  Arms: Spanish Version eBodyProject
Behavioral: Psychoeducationa Prevention Program — Participants in this group will receive a weekly newsletter with information about the beauty ideal, the costs of pursuing it, and tips for resisting the pressure to pursue this ideal, as well as tips for managing the emotions associated with it. However, they will not have to perform exercises related to this information, a psychoeducational intervention. Once the study is finished, these participants will receive an email again in case they are interested in taking part in the eBodyProject prevention program.
  Arms: Psychoeducational Prevention Program

SUMMARY:
The goal of this clinical trial is to analyze and compare in female college women two prevention programs for eating disorders, the Spanish Version of the eBodyProject and a traditional/educational prevention program. The main question it aims to answer is:

• The Spanish Version of the eBodyProject (intervention group) is more effective to prevent the onset of eating disorders with college students than a traditional psychological and educational prevention program (control group).

Participants will have to complete two main phases: assessment (pre- prevention program) and conducting the eBodyProject or traditional prevention program. The duration of the program is 4 weeks.

If there is a comparison group: Researchers will compare the Spanish eBodyProject Group with the traditional group to see and compare the effectiveness of each intervention arm.

DETAILED DESCRIPTION:
The main objective of this project is to validate the Spanish version of the eating disorder prevention program, eBodyProject, proving its effectiveness through its application in a female university population. A comparison will be made with a standard ACT reporting program.

The following specific objectives are proposed:

* Identify and analyze the risk factors for eating disorders in the university population
* Analyze the evolution of ED risk factors throughout the prevention program for each group (pre- and post-intervention).
* Analyze the differences between groups (eBodyProject vs. standard treatment) of the risk factors for eating disorders throughout the prevention program (pre- and post-intervention).
* Analyze long-term efficacy through follow-ups at 1, 3 and 6 months from the end of the program for both groups.
* Analyze adherence and satisfaction with the program.

What does the study involve?

eBodyProject Intervention

The Spanish adaptation of the eBodyProject program will be modified (Stice et al., 2012b). This program consists of 4 modules adapted from the most recent version of the original program The Body Project, presented by the original authors who have given their consent and suggestions for the realization of the Spanish version.

The activities proposed through the different modules will be in written format or behavioral activities aimed at criticizing the ideal of feminine beauty imposed by today's society and promoting self-acceptance. Specifically, each module pursues the following objectives:

* Module 1: Origin and definition of the ideal of beauty; Examine the costs of pursuing the beauty ideal
* Module 2: Explore and learn different ways of resisting pressure to pursue the ideal of beauty
* Module 3: Learning to manage and face our own concerns about appearance and cultural pressures on thinness
* Module 4: Learn new and more positive ways to talk about one's appearance Each module will be carried out independently, following the instructions provided in the web space. The time available to carry out each module will be one week, with an average duration of 40-45 minutes per module. Participants will receive feedback from the professional within the first 2-3 days after the completion of each module. For the promotion of participation, 1 day before the start of the module and 2 days before its completion will be remembered.

Psychoeducational intervention for group control

Participants in this group will receive a weekly newsletter with information about the beauty ideal, the costs of pursuing it, and tips for resisting the pressure to pursue this ideal, as well as tips for managing the emotions associated with it. However, they will not have to perform exercises related to this information, a psychoeducational intervention. Once the study is finished, these participants will receive an email again in case they are interested in taking part in the eBodyProject prevention program.

What are the possible benefits or risk for the participants?

Benefits

* Validation in a Spanish sample of a prevention program that has presented positive results in other countries for the university population. Therefore, the possibility of having a preventive tool for eating disorders and therefore reducing their prevalence among this population.
* Contribution in the field of ED prevention, both at the research and practice level. To have an effective and validated tool for the Spanish population.
* Reduction of intervention costs. Prove the efficacy in preventive programs have an impact on a lower prevalence of EDs and therefore less need for intervention. Reducing not only economic costs, but also reducing the personal costs resulting from suffering an eating disorder.
* Improve mental health in the university population that has been identified as a vulnerable population with high prevalence of psychological problems.

Risks This program is preventive and does not pose a risk to the physical or mental health of the participants. Following the inclusion and exclusion criteria, if serious cases of ED are detected, they will be referred to a more specialized treatment adapted to their needs.

If during the development of the program any participant reports discomfort or some type of negative repercussion, they will immediately be removed from the program and the case will be studied for referral if necessary.

Where is the study run from?

Spain

When is the study starting and how long is it expected to run for?

The study began on 1st November 2022, it is expecting to last two years.

Who is funding the study?

This study is not funded by any organization

Who is the main contact? Dra. Carmen Varela carmenvarela@ub.edu cvarela@ubu.es

ELIGIBILITY:
Inclusion Criteria:

1. Female college students
2. Currently studying college degree, master or post-degree
3. Participants must show inform consent
4. Age > 18 years

Exclusion Criteria:

1. Currently, absence of eating disorders or other several psychological problem
2. Currently on treatment for an eating disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Onset of Eating Disorders Symptomatology | 4 weeks
  Eating Attitudes Test -26 [EAT-26]

SECONDARY OUTCOMES:
State of Mood | 4 weeks
  Beck Depression Inventory [BDI]
Thin-ideal internalization | 4 weeks
  Sociocultural Attitudes Towards Appearance Questionnaire 4 [SATAQ-4]
Body Dissatisfaction | 4 weeks
  Body Shape Questionnaire [BSQ]
Eating Behaviors | 4 weeks
  The Dutch Eating Behavior Questionnaire [DEBQ]

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared to other researchers to ensure the anonymity of the participants.

REFERENCES:
- [Background] Stice E, Durant S, Rohde P, Shaw H. Effects of a prototype Internet dissonance-based eating disorder prevention program at 1- and 2-year follow-up. Health Psychol. 2014 Dec;33(12):1558-67. doi: 10.1037/hea0000090. Epub 2014 Jul 14. PMID 25020152
- [Background] Stice E, Onipede ZA, Marti CN. A meta-analytic review of trials that tested whether eating disorder prevention programs prevent eating disorder onset. Clin Psychol Rev. 2021 Jul;87:102046. doi: 10.1016/j.cpr.2021.102046. Epub 2021 May 21. PMID 34048952
- [Background] Stice, E., Rohde, P. & Shaw, H. (2013). The Body Project. Oxford.
- [Background] Stice E, Rohde P, Gau J, Shaw H. Effect of a dissonance-based prevention program on risk for eating disorder onset in the context of eating disorder risk factors. Prev Sci. 2012 Apr;13(2):129-39. doi: 10.1007/s11121-011-0251-4. PMID 21975593
- [Background] Stice E, Rohde P, Durant S, Shaw H. A preliminary trial of a prototype Internet dissonance-based eating disorder prevention program for young women with body image concerns. J Consult Clin Psychol. 2012 Oct;80(5):907-16. doi: 10.1037/a0028016. Epub 2012 Apr 16. PMID 22506791
- [Background] Luo YJ, Jackson T, Stice E, Chen H. Effectiveness of an Internet Dissonance-Based Eating Disorder Prevention Intervention Among Body-Dissatisfied Young Chinese Women. Behav Ther. 2021 Jan;52(1):221-233. doi: 10.1016/j.beth.2020.04.007. Epub 2020 Apr 19. PMID 33483119
- [Background] Beck, A. T., Steer, R. A. y Brown, G. (1996). Beck Depression Inventory-II (BDI-II). APA PsycTests. https://doi.org/10.1037/t00742-000
- [Background] Cebolla A, Barrada JR, van Strien T, Oliver E, Banos R. Validation of the Dutch Eating Behavior Questionnaire (DEBQ) in a sample of Spanish women. Appetite. 2014 Feb;73:58-64. doi: 10.1016/j.appet.2013.10.014. Epub 2013 Oct 28. PMID 24177441
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] Rivas T, Bersabe R, Jimenez M, Berrocal C. The Eating Attitudes Test (EAT-26): reliability and validity in Spanish female samples. Span J Psychol. 2010 Nov;13(2):1044-56. doi: 10.1017/s1138741600002687. PMID 20977051
- [Background] Sanz, J., Perdigón, A. L. y Vázquez, C. (2003). Adaptación española del Inventario para la Depresión de Beck-II (BDI-II): 2. Propiedades psicométricas en población general. Clínica y Salud, 14(3), 249-280. https://www.redalyc.org/pdf/1806/180617972001.pdf
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Van Strien T., Frijters J., Bergers G. y Defares P. (1986). The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional and external eating behaviors. International Journal of Eating Behaviors. https://doi.org/10.1002/1098108X(198602)5:2<295::AID-EAT2260050209>3.0.CO;2-